CLINICAL TRIAL: NCT06165224
Title: A Bidirectional Cohort Study of COMMD10 Expression in Tumor Tissues for Predicting Radiosensitivity
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-485
Record Dates: First submitted 2023-12-03; First posted 2023-12-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Biomarker; Radiosensitivity
Keywords: copper metabolism domain protein 10; biomarker; radiosensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — tumor tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiotherapy is one of the main treatments for malignant tumors, and according to authoritative estimates, about 70% of patients with malignant tumors should receive radiotherapy. However, radiation resistance limits its application and clinical curative effect. To find suitable radiation resistance markers and identify patients with radiation resistance, early part of the patients with appropriate radiotherapy sensitization agent or choose other more efficient and low toxicity of treatment, for improving the prognosis of patients, improve the quality of survival is of great significance, it is also the difficult point in the present study. However, there are no effective biomarkers to predict radiosensitivity. Through our previous basic research and analysis of clinical tumor tissues, we have found that the low expression of copper metabolism domain protein 10 (COMMD10) is associated with radioresistance, and COMMD10 is an effective marker for predicting radiosensitivity. We planned to conduct a single-center, prospective cohort study to verify the reliability of COMMD10 as a predictive marker for radiosensitivity in pan-cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old;
2. Voluntarily sign informed consent;
3. Nasopharyngeal carcinoma, head and neck tumor, lung cancer, breast cancer, stomach cancer, colorectal cancer, glioma, esophageal cancer, liver cancer, bile duct cancer, cervical cancer, prostate cancer confirmed by pathology;
4. Measurable tumor lesions according to RECIST v1.1 criteria;
5. Patients with radiation therapy indications and voluntarily accept radiotherapy;
6. ECOG PS score: 0/1.

Exclusion Criteria:

1. There are contraindications to radiotherapy;
2. Pathological sections could not be obtained;
3. Presence of metal metabolism-related diseases such as Wilson's disease;
4. Merge other tumors (has cured basal cell or squamous cell cancer, and cervical cancer in situ except 5);
5. Patients had any serious coexisting medical conditions that could pose an unacceptable risk or negatively affect trial adherence. "For example, unstable heart disease requiring treatment, chronic hepatitis, kidney disease, poor health status, uncontrolled diabetes (fasting blood glucose > 1.5 × ULN), and mental illness;"
6. The investigator judged that he was not suitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have solid tumor and need radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 month
  The objective response rate (ORR) is the proportion of patients who achieve a prespecified reduction in tumor volume that is maintained for a minimum duration. The objective response rate was defined as the sum of complete response plus partial response (CR+PR). According to RECIST1.1 criteria, CR was defined as the disappearance of target lesions and the reduction of the short diameter of pathological lymph nodes to less than 10mm. PR: the sum of the measured diameters of the target lesions reduced by 30% compared with the baseline; PD: the sum of the major diameters of all target lesions increased by at least 20%, and the absolute value of the sum of the major diameters increased by more than 5mm, or new lesions appeared. SD: Changes between PR and PD.

SECONDARY OUTCOMES:
Overall survival (OS) | 1 years
  OS was defined as the time from the date of inclusion until death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang hospital, Southern medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No